CLINICAL TRIAL: NCT06224023
Title: Predictive Values of Presepsin Levels in ASciteS in Patients With Chronic Liver Failure
Acronym: PASS
Status: Recruiting | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor of Gastroenterology, Carol Davila University of Medicine and Pharmacy
Other Study IDs: PASS
Record Dates: First submitted 2024-01-12; First posted 2024-01-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Ascites Hepatic; Liver Failure; Cirrhosis, Liver
MeSH Terms: conditions — Liver Failure; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ascites, peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic liver failure and ascites
  Interventions: Diagnostic Test: Determination of presepsin levels in ascites

INTERVENTIONS:
Diagnostic Test: Determination of presepsin levels in ascites — A diagnostic paracentesis will be performed and presepsin level will be determined in ascites.

SUMMARY:
The investigators aim to study the predictive value of presepsin in ascites in newly admitted patients with chronic liver failure.

DETAILED DESCRIPTION:
Presepsin is a plasmatic cleaved fragment of CD14. CD14 is a toll like receptor who has the role to identify certain lipopolysaccharides on the surface of bacteria (aerobes and anaerobes), thus promoting an inflammatory response.

A study of 153 patients with liver cirrhosis published by a team of investigators from Iasi, Romania, has proven an useful role of plasma presepsin in early diagnosis of infections in patients in acute on chronic liver failure.

In addition, plasma presepsin has been proposed as an independent predictor of mortality in patients with decompensated liver cirrhosis, without concomitant bacterial infections.

Question to be answered by this study The investigators aim to evaluate the predictive role of ascites presepsin in patients with chronic liver failure.

Hypothesis Presepsin levels in ascites may have a prognostic role in patients with ascites and chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* patient with ascites and chronic liver failure
* no contraindications and technical possibility to perform diagnostic paracentesis
* age above 18 years old
* informed consent

Exclusion Criteria:

* contraindications to paracentesis or technical impossibility to perform paracentesis
* absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted with chronic liver failure and ascites. A diagnostic paracentesis will be performed at the day of admission.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality at 6 months | 6 months
  Number of who deceased during admission or during the 180 days after admission divided by the number of patients who were admitted.
  An analysis will be done to see if the presepsin levels are predictive for this event.

SECONDARY OUTCOMES:
Spontaneous bacterial peritonitis (SBP) rate | 6 months
  The number of patients diagnosed with SBP during admission divided by the total number of patients. An analysis will be done to see if the presepsin levels are predictive for this event.
Hepatic encephalopathy rate | 6 months
  Number of patients diagnosed with hepatic encephalopathy during admission divided by the total number of patients.
  An analysis will be done to see if the presepsin levels are predictive for this event.
Any infection rate | 6 months
  The number of patients diagnosed with any infection during admission divided by the total number of patients.
  An analysis will be done to see if the presepsin levels are predictive for this event.

CONTACTS AND LOCATIONS:
Locations (1):
- "Agrippa Ionescu" Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Igna R, Girleanu I, Cojocariu C, Huiban L, Muzica C, Singeap AM, Sfarti C, Chiriac S, Petrea OC, Zenovia S, Nastasa R, Cuciureanu T, Stafie R, Stratina E, Rotaru A, Stanciu C, Blaj M, Trifan A. The Role of Presepsin and Procalcitonin in Early Diagnosis of Bacterial Infections in Cirrhotic Patients with Acute-on-Chronic Liver Failure. J Clin Med. 2022 Sep 15;11(18):5410. doi: 10.3390/jcm11185410. PMID 36143057
- [Background] Ferrarese A, Plebani M, Frigo AC, Burra P, Senzolo M. Presepsin as a biomarker of inflammation and prognosis in decompensated liver disease. J Hepatol. 2021 Jul;75(1):232-234. doi: 10.1016/j.jhep.2021.01.016. Epub 2021 Jan 21. No abstract available. PMID 33484772